CLINICAL TRIAL: NCT01873443
Title: An Open-Label, Single-Arm, Maintenance Study to Demonstrate Long-Term Efficacy and Safety of CT-P10 in Patients With Rheumatoid Arthritis Who Were Treated With Rituximab (MabThera or CT-P10) in Study CT-P10 1.1
Brief Title: Long-Term Efficacy and Safety of CT-P10 in Patients With RA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P10 1.3; 2012-005502-21 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-06-10 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab, MTX, folic acid (Experimental)
  Interventions: Drug: Rituximab, MTX, folic acid

INTERVENTIONS:
Drug: Rituximab, MTX, folic acid — Rituximab IV 1000mg MTX 10~25mg/week Folic acid at least 5mg/week
  Other Names: Rituximab=CT-P10

SUMMARY:
This is an open-label, single-arm, multicenter, efficacy, and safety maintenance study of the Phase 1 Study CT-P10 1.1. This study is designed to assess the long-term efficacy and safety of CT-P10 co-administered with MTX and folic acid in patients with RA who have completed the scheduled visits in Study CT-P10 1.1

ELIGIBILITY:
Inclusion Criteria:

* Patient has disease improvement (moderate or good response) according to Disease Activity Score using 28 joint counts (DAS28) during the last course of treatment in Study CT-P10 1.1.
* Patient has completed all of the scheduled visits in the Study CT-P10 1.1 Main Study Period, including the Core Study Period and/or Extension Study Period.

Exclusion Criteria:

* Patient has been withdrawn from Study CT-P10 1.1 for any reason.
* Patient has, at the time of providing informed consent, any current medical issues such as serious adverse events (SAEs) or current or previous intolerance issues that mean continuation in this maintenance study could be detrimental to their health, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation by ACR criteria and safety evaluation by hypersensitivity monitoring | 8 week interval
  Efficacy will be assessed by evaluation of ACR criteria (ACR 20% , ACR 50% , ACR 70%, and hybrid ACR response), Safety will be assessed by evaluation of hypersensitivity monitoring via vital sign measurements (including blood pressure, heart and respiratory rates, and body temperature),etc,.

CONTACTS AND LOCATIONS:
Overall Officials: DaeHyun Yoo, Ph.D, Study Director — Hanyang University
Locations (1):
- Inha University College of Medicine Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Park W, Suh CH, Shim SC, Molina FFC, Jeka S, Medina-Rodriguez FG, Hrycaj P, Wiland P, Lee EY, Shesternya P, Kovalenko V, Myasoutova L, Stanislav M, Radominski S, Lim MJ, Choe JY, Lee SJ, Lee SY, Kim SH, Yoo DH. Efficacy and Safety of Switching from Innovator Rituximab to Biosimilar CT-P10 Compared with Continued Treatment with CT-P10: Results of a 56-Week Open-Label Study in Patients with Rheumatoid Arthritis. BioDrugs. 2017 Aug;31(4):369-377. doi: 10.1007/s40259-017-0233-6. PMID 28600696